CLINICAL TRIAL: NCT00322764
Title: Dose-Escalating, Phase II Study to Assess the Safety and Tolerability of RG2417 in the Treatment of Bipolar I Depression
Brief Title: Phase II Study to Assess RG2417 in the Treatment of Bipolar I Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repligen Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RG2417-01
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-11

CONDITIONS: Bipolar Depression
Keywords: manic depression; bipolar disorder; depression; uridine; RG2417
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Uridine

INTERVENTIONS:
Drug: Uridine

SUMMARY:
The primary purpose of this study is to determine the safety and efficacy of oral RG2417 (Uridine) when administered to patients with Bipolar I depression twice daily for six weeks.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV-TR diagnosis of Bipolar I Depression
2. 18 to 65 years of age, inclusive
3. Depressive phase, as measured by MADRS greater than or equal to 20 at Screening and Day1
4. Duration of current depressive episode of at least four weeks by Day 1
5. Competent to give informed consent

Exclusion Criteria:

1. Manic/hypomanic/mixed episode as determined by the MINI at Screening and/or a Young Mania Rating Scale (YMRS) score of > 12 at Screening and/or Day 1
2. Dementia or any current Axis I diagnosis (excluding bipolar I) requiring pharmacological treatments
3. A history of alcohol or substance dependence within six months of Day 1, or a history of alcohol or substance abuse within three months of Day 1
4. Urine drug screen positive for amphetamines, cocaine metabolites, opiates and/or phencyclindine (PCP)
5. An Axis II diagnosis that is likely to interfere with protocol compliance
6. Initiation of or increase in psychotherapy within 4 weeks of Screening
7. Psychotropic medication (excluding fluoxetine) within 24 hours of initiation of study drug on Day 1; fluoxetine within 2 weeks of initiation of study drug on Day 1
8. Serious suicidal or homicidal risk as determined by the investigator and/or a score of > 5 on the suicide item #10 of the MADRS at Screening and/or Day 1
9. History of sensitivity to any of the ingredients in the study drug
10. Clinically significant abnormality in any screening laboratory results
11. Clinically significant organic disease, including cardiovascular, endocrine, hepatic, pulmonary, neurologic, or renal disease, or any other medical condition, serious intercurrent illness, or extenuating circumstances that, in the opinion of the investigator, would interfere with the performance or interpretability of, or put the patient at risk from, the study procedures
12. Women who are pregnant, breastfeeding, or refuse to use adequate birth control
13. Current seizure disorder
14. Participation in an investigational drug study within twenty-eight days of Day 1
15. Current psychotic episode
16. Clozaril use and/or electroconvulsive therapy within six months of Day 1
17. Failure of three or more adequate trials of standard therapies for depression during the current episode
18. Current episode of depression is longer than one year

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-03

PRIMARY OUTCOMES:
Improvement of MADRS and CGI BP C for RG2417 treatment in comparison to placebo

CONTACTS AND LOCATIONS:
Overall Officials: David Jacoby, MD, PhD, Study Director — Repligen Corporation
Locations (11):
- United States (11):
  - Stanford University, Stanford, California
  - Carman Research, Smyrna, Georgia
  - Indiana University-Purdue University Indianapolis, Indianapolis, Indiana
  - Marc Hertzman, MD, PC, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Medical & Behavioral Health Research, PC, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Future Search Trials of Austin, Austin, Texas
  - Future Search Trials of Dallas, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas